CLINICAL TRIAL: NCT00006087
Title: A Randomized Prospective Study Comparing Annual Chest X-Rays to Annual Spiral Chest CT Scanning in Patients at High-Risk for the Development of Lung Cancer
Brief Title: Chest X-Ray or Chest CT Scan in Patients at High Risk of Developing Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jewish Hospital and St. Mary's Healthcare (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000068079; JHL-45199; NCI-V00-1600
Record Dates: First submitted 2000-08-03; First posted 2003-12-23 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-12

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — X-Rays

INTERVENTIONS:
Procedure: annual screening
Procedure: bronchoscopic and lung imaging studies
Procedure: comparison of screening methods
Procedure: computed tomography
Procedure: radiography
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Diagnostic procedures such as chest x-ray and chest CT scans may be effective in early detection of lung cancer.

PURPOSE: Randomized clinical trial to compare the effectiveness of a chest CT scan given once a year with that of a chest x-ray given once a year in detecting lung cancer in patients at a high-risk of developing lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of a lung cancer risk assessment questionnaire combined with spirometry testing in identifying a statistically significant number of persons with high-risk behaviors for the development of lung cancer. II. Determine the sensitivity of these screening techniques in identifying a population at high risk for the development of lung cancer. III. Determine the number of patients necessary to screen in order to identify the high-risk population eligible for this study. IV. Determine the lead time bias of CT scans versus chest x-rays in these patients. V. Determine the efficacy of spiral CT scanning of the chest in detecting early lung cancers not visible on chest x-rays in patients at high risk for lung cancer. VI. Compare annual spiral CT scanning versus annual chest x-rays in detecting lung cancer in these patients. VII. Compare survival and fatality in these patients with these detection methods.

OUTLINE: Patients are randomized to one of two screening arms. Arm I: Patients receive routine medical care, an annual nursing assessment, and an annual chest x-ray. Any new abnormality identified is further evaluated through standard acceptable medical interventions. Arm II: Patients receive routine medical care, an annual nursing assessment, and an annual spiral CT scan of the chest. If an abnormal mass greater than 10 mm in diameter or 5-10 mm in diameter and highly suspicious for malignancy is detected, chest x-ray and tissue diagnosis is obtained. If the abnormal mass is 10 mm or less in diameter, a thin section high resolution image of the mass is obtained. If this image is normal or benign, annual spiral CT scanning is continued. If the image is indeterminate, a repeat high resolution scan is performed in 3 months. If the image is unchanged at 3 months, annual spiral CT scanning is continued. If the mass is larger at 3 months, chest x-ray and tissue diagnosis is performed. Screening continues for 5 years in the absence of disease detection.

PROJECTED ACCRUAL: A minimum of 1,000 patients (500 per screening arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients at high risk for the development of lung cancer as defined by the following: At least 40 pack years smoking (may have stopped smoking within past 10 years) at time of study entry FEV-1/FVC ratio less than 70% predicted OR FEV-1 less than 80% predicted obtained from 3 serial performances with less than 5% difference Normal or stable current chest x-ray

PATIENT CHARACTERISTICS: Age: 40 to 70 Performance status: Not specified Life expectancy: At least 5 years Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Pulmonary: See Disease Characteristics Other: No other comorbidity that limits life span to less than 5 years No prior cancer except nonmelanomatous skin cancer or carcinoma in situ of the cervix Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, FACP, Study Chair — Kentuckiana Cancer Institute, PLLC
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States